CLINICAL TRIAL: NCT00062075
Title: A Phase 2 Study of Depsipeptide in Patients With Relapsed or Refractory AML
Brief Title: Romidepsin in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00034; 12209B; CDR0000304460; N01CM62201 (NIH); N01CM17102 (NIH); U01CA099177 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-04

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Leukemia, Myeloid, Acute | interventions — romidepsin

ARMS (1):
- Treatment (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax

SUMMARY:
This phase II trial is studying how well romidepsin works in treating patients with relapsed or refractory acute myeloid leukemia. Drugs used in chemotherapy, such as romidepsin, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the complete and partial response rate in patients with relapsed or refractory acute myeloid leukemia treated with FR901228 (depsipeptide).

II. Determine the toxicity of this drug in these patients. III. Correlate clinical response with specific cytogenetic abnormalities in patients treated with this drug.

OUTLINE: Patients are stratified according to the presence of a specific chromosomal abnormality (t[8;21] vs inv 16 vs t[15;17] vs absence of these chromosomal abnormalities).

Patients receive romidepsin IV over 4 hours on days 1, 8, and 15.

Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed acute myeloid leukemia (AML) defined by the WHO classification
* Initial diagnosis with either of the following:

  * Bone marrow or peripheral blood myeloblasts of at least 20%,
  * Recurring genetic abnormalities (e.g., t[8;21], inv 16, or t[16;16]) and
  * Bone marrow blast percentage less than 20%
* Relapsed or refractory disease defined by 1 of the following:

  * Under 60 years of age and in second relapse or greater,
  * Over 60 years of age and in first relapse,
  * Acute promyelocytic leukemia that has relapsed despite prior tretinoin and arsenic therapy,
  * Primary refractory AML for which no standard therapy exists
* Patients who are over 60 years of age with previously untreated disease and who refuse conventional chemotherapy are eligible
* Patients who are over 60 years of age and in first relapse and poor medical candidates for reinduction chemotherapy or who refuse conventional chemotherapy are eligible
* Not medically appropriate for OR refused curative bone marrow or stem cell transplantation
* No CNS leukemia
* ECOG 0-2 OR Karnofsky 60-100%
* LVEF at least 40% by MUGA
* QTc interval less than 500 msec by EKG
* No myocardial infarction within the past 3 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to FR901228 (depsipeptide)
* No concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection
* At least 4 weeks since prior autologous stem cell or bone marrow transplantation
* No prior allogeneic stem cell or bone marrow transplantation
* No concurrent biologic agents
* At least 2 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas)
* No concurrent chemotherapy, concurrent hydroxyurea allowed during the first course of study therapy to control hyperleukocytosis
* No concurrent radiotherapy
* Recovered from prior therapy
* At least 4 weeks since prior investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No concurrent drugs known to have histone deacetylase inhibitor activity (e.g., sodium valproate)
* No other concurrent antineoplastic agents
* No prior FR901228 (depsipeptide)
* At least 2 weeks since prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2003-05; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial) | Up to 7 years
Adverse events, measured using National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 2.0 | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Vanderbilt University, Nashville, Tennessee